CLINICAL TRIAL: NCT06542042
Title: Application of Oxford Nanopore Adaptive Sequencing Method in Infection Post Liver Transplantation
Brief Title: Application of Nanopore Adaptive Sequencing
Status: Not yet recruiting | Type: Observational
Sponsor: Shenzhen Third People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SZSY001; 2022YFC2304700 (Other Grant/Funding Number: Ministry of Science and Technology)
Record Dates: First submitted 2024-06-27; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-06

CONDITIONS: Liver Transplant Infection
Keywords: Oxford nanopore adaptive sequencing method

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NAS group: In this group, the investigators will detect the number of pathogen in alveolar lavage fluid, blood and peritoneal drainage by using NAS.
  Interventions: Diagnostic Test: NAS, NGS and Laboratory tests
- NGS group: In this group, the investigators will detect the number of pathogen in alveolar lavage fluid, blood and peritoneal drainage by using NGS.
  Interventions: Diagnostic Test: NAS, NGS and Laboratory tests
- Lab Tests group: In this group, the investigators will detect the number of pathogen in alveolar lavage fluid, blood and peritoneal drainage by using laboratory tests.
  Interventions: Diagnostic Test: NAS, NGS and Laboratory tests

INTERVENTIONS:
Diagnostic Test: NAS, NGS and Laboratory tests — Using three diffrent detection methods and comparing their efficiency

SUMMARY:
Infection post liver transplantation is an important factor in the death in patients. The traditional method of diagnosing infection post liver transplantation is laboratory tests. But the sensitivity and specificity of blood tests is poor. Next-generation sequencing (NGS) has greater detection rate for mycobacterium tuberculosis, anaerobes and fungi and greater sensitivity compare with blood tests. However use of NGS is limited because of the short read-length. Oxford nanopore adaptive sequencing (NAS) method is the Third Revolution in Sequencing Technology. For each 1 Gbp of data, NAS sequencing detected 45 times more microbiome sequences than Nanopore standard sequencing and 2.5 times more than Illumina sequencing. The purpose of this study is to compare NAS with NGS and laboratory tests for the diagnostic rate of infection post liver transplantation.

DETAILED DESCRIPTION:
Based on the previous work, the investigators found that: 1. NAS has a higher microbial enrichment efficiency and can detect pathogenic information more quickly compared with nanopores normal sequencing (NNS); 2. NAS can detect more specific pathogen fragments with short-time sequencing; 3. NAS can cover more pathogenic genomes than NNS in a short-time; 4. NAS can detect antibiotic resistance information of pathogenic bacteria in clinical samples.

ELIGIBILITY:
Inclusion Criteria:

* Accept liver transplantation
* Signing informed consent voluntarily
* Possessing ability to comprehend material information
* Participating this study voluntarily

Exclusion Criteria:

* Participated another study
* Graft loss
* Have undergone a multi-organ transplantion or have had a previous organ transplantation
* Patient died

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited randomly and if they violate the protocol or occur clinical adverse events, the investigators will ask them to withdraw from this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosed infection post liver transplantation | Post liver transplantation before patients discharge from hospital, an average of 1 months.
  Any pathogens are detected in alveolar lavage fluid, peritoneal drainage or blood before patients discharge from hospital, an average of 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zhong, Dr, Principal Investigator — Shenzhen Third People's Hospital
Locations (1):
- Shenzhen Third People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheng H, Sun Y, Yang Q, Deng M, Yu Z, Zhu G, Qu J, Liu L, Yang L, Xia Y. A rapid bacterial pathogen and antimicrobial resistance diagnosis workflow using Oxford nanopore adaptive sequencing method. Brief Bioinform. 2022 Nov 19;23(6):bbac453. doi: 10.1093/bib/bbac453. PMID 36259361